CLINICAL TRIAL: NCT05068323
Title: Impact of Interictal Epileptiform Activity on Some Cognitive Domains in Newly Diagnosed Epileptic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shady Mohamed Safwat Hassan, Lecturer of Neurology, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Epilepsy and Cognition
Record Dates: First submitted 2021-09-20; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Impairment; Epilepsy
MeSH Terms: conditions — Cognitive Dysfunction; Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: case control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epilepsy (Other): Newly diagnosed epileptic patients
  Interventions: Diagnostic Test: Digital electroencephalography (EEG) for an hour (16 channels)
- Control (Sham Comparator): healthy subjects
  Interventions: Diagnostic Test: Digital electroencephalography (EEG) for an hour (16 channels)

INTERVENTIONS:
Diagnostic Test: Digital electroencephalography (EEG) for an hour (16 channels) — Digital electroencephalography (EEG) for an hour (16 channels)

SUMMARY:
Epilepsy is a common health problem worldwide. In general population, studies in developed countries estimated the annual incidence of epilepsy to be~50 per 100,000 and prevalence to be ~8.2 per 1,000. These figures are higher in developing countries in which prevalence of >10 per 1,000 was reported. In Upper Egypt, Assiut Governorate, the prevalence rate was 12.9 per 1,000.

In people with epilepsy there is an associated high rate of cognitive difficulties that compromise educational progress and achievement throughout life. Approximately 1-5% of the population exhibits epileptiform discharges on electroencephalography (EEG). Interictal epileptiform discharges (IEDs), meaning spikes, polyspikes, sharp waves, or spike and slow-wave complexes without observed clinical seizures, are commonly observed in patients with epilepsy.

Epilepsy syndromes manifesting with IEDs are detrimental to cognitive function. Recently, two studies found that frequent IEDs can impair cognitive performance in children. and adult patients. Several studies indicated that IEDs in patients with epilepsy had a disruptive effect on information processing speed with even a low percentage of IEDs (1%).However, it is unclear whether IEDs are associated with disrupted academic performance in patients with idiopathic epilepsy, and the relationship between general cognitive ability and academic performance in those patients has not been clarified.

Understanding how IEDs interfere with neurocognitive outcomes is important ,while the goal of medical and surgical treatments for epilepsy is to achieve seizure-freedom with minimal morbidity, the benefits of IED suppression are more controversial.

DETAILED DESCRIPTION:
This study aims to

1. Evaluate the influence of interictal epileptiform activity per se on some cognitive functions in newly diagnosed patients with epilepsy (before using anti-seizure medications)
2. Determine different effects among different brain areas (producing epileptiform activity) on specific cognitive domains Type of the study: Case control Study Study Setting: Assiut university hospital -Neuropsychiatry hospital- Out patient clinics.

Study subjects: Will include epilepsy patients that diagnosed according to the International League Against Epilepsy criteria, 2017:

Study tools All patients included in this study will be subjected to: -

1. History taking including Personal history, history of present illness, therapeutic history, past history and family history
2. Complete physical examination. 3) Neurological examination. 4) Digital electroencephalography (EEG) for an hour (16 channels). 5) Psychiatric assessment: all subjects included in the study will be asked to perform a series of psychological tests done by expert psychologist to detect cognitive impairment

   1. Montreal Cognitive Assessment(MoCA).
   2. Hamilton Depression Rating Scale (HDRS).

ELIGIBILITY:
Inclusion Criteria:

- a) Patients [with age ranges from 10 to 50 years] of both sex. b) Patients with confirmed diagnosis of idiopathic localization-related or generalized epilepsy.

c) Either before receiving anti-epileptic drugs or on regular treatment with antiepileptic drugs for less three months.

Exclusion Criteria:

1. Patients with symptomatic or secondary epilepsies either due to general medical conditions or drug induced.
2. Other neurological , psychiatric or metabolic disorders that affect cognition.
3. Regular use of antiepileptic medications more than three months.
4. utilization of regular medications other than AEDs that affect cognition.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of some High frequency epileptiform discharges measured by HZ on some cognitive domines using electroencephalogram | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shady Mohamed Safwat Mohamed Tawfik Hassan, Asyut, Egypt